CLINICAL TRIAL: NCT04137900
Title: A First-in-Human, Multicenter, Open-Label, Phase 1 Dose-Escalation and Cohort Expansion Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAB004 as Monotherapy and in Combination With Toripalimabin Subjects With Advanced Solid Malignancies Including Lymphoma
Brief Title: Safety, Tolerability and Pharmacokinetics of a Monoclonal Antibody Specific to B-and T-Lymphocyte Attenuator (BTLA) as Monotherapy and in Combination With an Anti-PD1 Monoclonal Antibody for Injection in Subjects With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TopAlliance Biosciences (Industry)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other); CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAB004-01
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Advanced Unresectable Solid Tumor; Metastatic Solid Tumor
Keywords: immunotherapy; BTLA; HVEM; check point inhibitor; solid tumor; non-small cell lung cancer; NSCLC; melanoma; lymphoma; monoclonal antibody; phase 1 trial
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Melanoma; Lymphoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- TAB004 0.3 mg/kg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004
- TAB004 1 mg/kg repeat dose every 21days up to 2 years (Experimental)
  Interventions: Drug: TAB004
- TAB004 3 mg/kg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004
- TAB004 10 mg/kg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004
- TAB004 200mg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004
- TAB004 20mg and Torpalimab 240mg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004; Drug: Toripalimab
- TAB004 70mg and Torpalimab 240mg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004; Drug: Toripalimab
- TAB004 200mg and Torpalimab 240mg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004; Drug: Toripalimab
- TAB004 500mg and Torpalimab 240mg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Drug: TAB004; Drug: Toripalimab

INTERVENTIONS:
Drug: TAB004 — Recombinant humanized IgG4κ monoclonal antibody specific to BTLA for injection
  Other Names: JS004
Drug: Toripalimab — a human IgG4k monoclonal antibody that specifically binds to the programmed death 1 (PD-1)
  Other Names: TAB001; JS001
  Arms: TAB004 200mg and Torpalimab 240mg repeat dose every 21 days up to 2 years; TAB004 20mg and Torpalimab 240mg repeat dose every 21 days up to 2 years; TAB004 500mg and Torpalimab 240mg repeat dose every 21 days up to 2 years; TAB004 70mg and Torpalimab 240mg repeat dose every 21 days up to 2 years

SUMMARY:
The primary objective is to assess the safety and tolerability of TAB004 as monotherapy and in combination with toripalimab in subjects with selected advanced solid malignancies, including lymphoma, and to evaluate the recommended Phase 2 dose.

The secondary objectives are to: 1) describe the pharmacokinetic (PK) profile of TAB004 monotherapy and in combination with toripalimab and to describe the PK profile of toripalimab when administered with TAB004, 2) evaluate antitumor activity of TAB004 monotherapy and in combination with toripalimab; and 3) determine the immunogenicity of TAB004 monotherapy and in combination with toripalimab and to determine the immunogenicity of toripalimab when administered with TAB004.

The exploratory objectives are to: 1) evaluate pharmacodynamic effects of TAB004 on its target receptor BTLA, as well as effects on the immune system; 2) evaluate biomarkers that may correlate with activity of TAB004 as monotherapy and in combination with toripalimab; 3) evaluate the utility of BTLA ligand, herpesvirus-entry mediator (HVEM), and additional exploratory biomarkers that could aid in selection of appropriate subjects for TAB004 monotherapy and in combination with toripalimab.

DETAILED DESCRIPTION:
OVERVIEW: This is a Phase 1, multi-center, open-label, dose-escalation study of TAB004, a recombinant humanized IgG4κ monoclonal antibody specific to BTLA when administered alone and in combination with toripalimab, a human IgG4k monocloncal antibody that specifically binds to the programmed death 1 (PD-1). It is estimated that up to 499 subjects with selected advanced solid malignancies (i.e.; non-small cell lung cancer [NSCLC], melanoma, renal cell carcinoma (RCC), urothelial carcinoma (UC), or other tumors), including lymphoma will be enrolled in the study.

Subjects must have a histologically or cytologically confirmed advanced unresectable or metastatic solid tumor, including lymphoma.

The study has 4 parts; Part A dose-escalation, Part B cohort expansion, Part C dose-escalation and Part D cohort expansion. In Part A, up to 24 subjects will be enrolled who must have received, or be ineligible for, or intolerant of, all available approved or standard therapies know to confer clinical benefit including immunotherapy, or for whom no standard therapy exists.

In Part B, C and D, subjects must have received at least one line of therapy for advanced or metastatic disease, but are not required to have received all standard therapies known to confer clinical benefit.

Part A is the monotherapy dose-escalation portion of the study. Four TAB004 dose levels are planned and include: 0.3, 1, 3 and 10 mg/kg. Part A will be the traditional 3 + 3 design with 3 to 6 subjects per dose level (cohort) and will receive their assigned dose every 21 days in the absence of a dose limiting toxicity (DLT) that would prevent further dosing.

Part B is the monotherapy cohort expansion portion of the study and will consist of up to 50 subjects in each advanced solid tumor indication (up to 200 subjects) that may include but not be limited to lymphoma, melanoma, NSCLC, or other tumors with agreement of the Sponsor.

Part C is the combination therapy dose-escalation portion of the study. Four dose levels are planned as follows: Cohort 1 - TAB004 20 mg and toripalimab 240mg; Cohort 2 - TAB004 70 mg and toripalimab 240 mg; Cohort 3 -TAB004 200 mg and toripalimab 240 mg; Cohort 4- TAB004 500 mg and toripalimab 240 mg. Part C will be the traditional 3 + 3 design with 3 to 6 subjects per dose level (cohort) and will receive their assigned doses every 21 days in the absence of a DLT that would prevent further dosing.

Part D is the combination therapy cohort expansion portion of the study. Up to 50 subjects will be enrolled in each advanced solid tumor indication (melanoma, NSCLC, RCC, UC, lymphoma) (up to 250 subjects). Doses of TAB004 and toripalimab will be determined based upon safety and efficacy data from Part C.

Tumor response will be evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1), the immune-related Response Evaluation Criteria in Solid Tumors (irRECIST), or the New Response Evaluation Criteria in Lymphoma (RECIL) 2017.

In the absence of confirmed disease progression and intolerable toxicities, subjects will be allowed to continue TAB004 (Part A and B) or TAB004 and toripalimab (Part C and D) administration every 21 days for up to 2 years.

DOSAGE AND ADMINISTRATION TAB004 doses are 0.3, 1, 3, 10 mg/kg, 20mg, 70mg, 200mg and 500mg. Toripalimab dose is 240mg. TAB004 alone or TAB004 plus toripalimab will be administered as a 60-minute i.v. infusion for the first dose and may be decreased at the investigators discretion to 30 minutes in subsequent infusions.

SAFETY EVALUATIONS Assessment of safety will be determined by vital sign measurements, clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status evaluations, diagnostic imaging, physical examinations, electrocardiograms, and the incidence and severity of adverse events.

Safety will also include evaluations of immune safety and immunogenicity. Blockade of BTLA pathway and PD-1 pathway by monoclonal antibodies has been demonstrated in several syngeneic mouse models to enhance specific T cell responses and inhibit tumor growth. In studies of BTLA deficient mice, diseases such as asthma, autoimmune involvement of the central nervous system, and systemic lupus erythematosus were exacerbated. Particular attention will be given to symptoms related to those diseases. The occurrence of adverse events that may follow enhanced T-cell activation such as pneumonitis, colitis, nephritis, severe skin reactions, endocrinopathies, or other immune-related adverse events (irAEs) will be evaluated for subjects receiving TAB004 alone or in combination with toripalimab.

An irAE is a clinically significant adverse event of any organ that is associated with drug exposure, of unknown etiology, and is consistent with an immune-mediated mechanism.

EFFICACY EVALUATIONS will include best overall response, objective response rate, duration of response or duration of stable disease, progression free survival and overall response.

PHARMACOKINETIC EVALUATIONS Pharmacokinetic parameters include AUC0-inf, AUC0-last, AUC0-21d, Cmax, Cmin trough, Tmax, t1/2, CL, accumulation and Vss.

STATISTICAL METHODS Part A and Part C are based on the 3+3 design for dose escalation and safety evaluation requirements. In Part B and Part D, sample size is estimated using Simon's two-phase design minimax method.

All PK/Pharmacodynamic, immunogenicity, and safety data will be summarized and presented by cohort as well as overall for the study, using descriptive statistics (number of subjects, mean, median, standard deviation, minimum, and maximum) for continuous variables and using frequencies and percentages for discrete variables.

ORR and the associated 2-sided 95% exact confidence limits will be calculated. The proportion of subjects who have experienced best response as CR, PR, SD, or progressive disease (PD) will be provided by cohorts in Part B and Part D.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and willing to sign the Informed Consent Form;
* 2. Male or female ≥ 18 years;
* 3. Subjects with histologically or cytologically confirmed advanced unresectable or metastatic solid tumor, including lymphoma that have progressed following prior treatment. In Part A, subjects must have received, or be ineligible for or intolerant of all available approved or standard therapies known to confer clinical benefit including immunotherapy, or for whom no standard therapy exists; in Part B, subjects with advanced or metastatic solid tumors, including but not limited to lymphoma, melanoma, NSCLC, or other tumors with agreement of the Sponsor, who must have received at least one line of therapy for advanced or metastatic disease, but are not required to have received all standard therapies known to confer clinical benefit; In Part C, subjects must have received at least one line of therapy for advanced or metastatic disease but are not required to have received all standard therapies known to confer clinical benefit; In Part D, subjects with advanced or metastatic solid tumors that may include but not limited to lymphoma, melanoma, NSCLC, RCC or UC who must have received at least one line of therapy for advanced or metastatic disease, but are not required to have received all standard therapies known to confer clinical benefit.
* 4. Measurable disease per RECISTv1.1 and iRECIST, or RECIL 2017 for lymphoma
* 5. ECOG performance status of 0 or 1 with life expectancy of 3 months in the opinion of the investigator.
* 6. Adequate organ and marrow function, as defined below:

  1. Hemoglobin 8.0 g/dL within first 2 weeks prior to first dose of TAB004 (are not requiring a transfusion within 14 days prior to dosing)
  2. Absolute neutrophil count (ANC) 1.0 x 109 /L (1,000 /mm3)
  3. Absolute lymphocyte count ≥ 0.6 x 109/L (600/mm3)
  4. Platelet count 75 x 109 /L (75,000 /mm3), and not requiring platelet transfusions within the 5 days prior to dosing
  5. Total bilirubin ≤ 1.5 x ULN except subjects with documented Gilbert's syndrome who must have a baseline total bilirubin ≤ 3.0 mg/dL
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN; for subjects with hepatic metastases, ALT and AST ≤ 5 x ULN
  7. Serum creatinine ≤ 1.5 x ULN OR calculated creatinine clearance (CrCl) or 24 hour urine CrCl ≥ 40 mL/minute Cockcroft-Gault formula will be used to calculate CrCl. 24-hour urine CrCl will be derived using the measured creatinine clearance formula
  8. International normalized ratio (INR) ≤ 2.0 and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN; applies only to subjects who do not receive therapeutic anticoagulation; subjects receiving therapeutic anticoagulation (such as low-molecular weight heparin or warfarin) should be on a stable dose
* 7. Willingness to provide consent for biopsy samples (In Part A, fresh pre-treatment biopsies will be requested from subjects with safely accessible lesions. For subjects who cannot provide a fresh pre-treatment biopsy, request for the most recent accessible archival specimen will be required. In Part B, C and D, fresh pre-treatment biopsies will be required from subjects with safely accessible lesions. The most recent archival specimens will also be requested).
* 8. Females of childbearing potential who are sexually active with a nonsterilized male partner must use effective contraception from time of screening, and must agree to continue using such precautions for 90 days after the final dose of TAB004 or toripalimab; cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
* 9. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as at least 12 months with no menses confirmed by follicle-stimulating hormone [FSH] levels. FSH testing will be conducted at the Screening visit to confirm post-menopausal status).
* 10. Subjects must use effective contraception. Nonsterilized males who are sexually active with a female partner of childbearing potential must use effective contraception from Day 1 and for 90 days after receipt of the final dose of TAB004 or toripalimab.

Exclusion Criteria:

* 1. Concurrent enrollment in another clinical study, unless it is an observational (non interventional) clinical study or the follow-up period of an interventional study.
* 2. Any concurrent anti-cancer therapy, such as but not limited to chemotherapy, targeted therapy, radiotherapy, immunotherapy, or biologic therapy. Radiation treatment for palliative intent is allowed provided that lesions other than those receiving radiation are available to measure response. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for type 2 diabetes and hormone replacement therapy) is acceptable.

Note: Local treatment of isolated lesions for palliative intent is acceptable (e.g., by local surgery or radiotherapy).

* 3. Receipt of any investigational anticancer therapy within 28 days prior to the first dose of TAB004 or, provided documentable, 5 half lives whichever is shorter, except for lymphoma in which the exclusionary period is 2 weeks for immune checkpoint inhibitors only.
* 4. Current or prior use of immunosuppressive medication within 2 weeks prior to the first dose of TAB004, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids not to exceed 10 mg/day of prednisone or equivalent.
* 5. Prior exposure to anti-BTLA, or anti-HVEM antibodies for subjects enrolled into Part A and B only; prior treatment with anti-PD-1 or anti-PDL-1is allowed,including toripalimab for all subjects.
* 6. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* 7. Subjects with another malignancy, or history or other malignancy within 3 years that is not expected to relapse. Subjects with non-melanomatous skin cancer or cervical cancer that has been curatively surgically resected are eligible.
* 8. Major surgery (as defined by the investigator) within 28 days prior to first dose of TAB004 or has not recovered to at least Grade 1 from adverse effects from such procedure, or anticipation of the need for major surgery during study treatment.
* 9. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to baseline or to NCI-CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of neuropathies that are stable or improving and alopecia. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by TAB004 may be included (e.g., hearing loss) after consultation with the medical monitor.
* 10. Active or prior documented autoimmune disease, such as but not limited to systemic lupus erythematosus, multiple sclerosis, inflammatory bowel diseases, rheumatoid arthritis, autoimmune hepatitis, systemic sclerosis, autoimmune vasculitis, autoimmune neuropathies or type 1 insulin-dependent diabetes mellitus.

Note: Subjects with the following are not excluded: vitiligo; alopecia; Grave's disease not requiring systemic treatment other than thyroid hormone replacement (within the past 2 years) psoriasis not requiring systemic treatment; controlled celiac disease; subjects with a history of autoimmune hypothyroidism requiring only thyroid hormone replacement therapy; And type 2 diabetes, provided that it is adequately controlled.

* 11. Clinically significant (intracranial, gastrointestinal) bleeding within 2 weeks prior to screening.
* 12. Known history of tuberculosis.
* 13. Subjects with history of or current drug-induced interstitial lung disease or pneumonitis ≥ Grade 2.
* 14. Subjects who have discontinued prior immune therapy due to immune mediated adverse reaction(s).
* 15. Subjects who are known to be human immunodeficiency virus positive.
* 16. Subjects with evidence of hepatitis B or C virus infection, unless their hepatitis is considered to have been cured. (Note that subjects with prior hepatitis B virus infection must have HBV viral load < 100 IU/mL before study enrollment, and must be treated according to local standards; hepatitis C virus infection must have, before study enrollment, no detectable viral load and must be treated according to local standards).
* 17. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis). Infection-related bowel inflammation, such as Clostridium difficile colitis, is not excluded provided that it has been fully resolved for ≥ 6 weeks.
* 18. History of anaphylaxis, or eczema that cannot be controlled with topical corticosteroids asthma.
* 19. Adult asthma that is moderate or severe, or asthma that has required: hospitalization in the last 2 years; invasive mechanical ventilation ever; systemic corticosteroids in the past year for exacerbations; or more than two short acting beta agonist (e.g., albuterol) administrations per month for breakthrough asthma symptoms. A history of childhood asthma or the presence of mild adult asthma that at baseline has symptoms that can be controlled well with inhaled corticosteroids or short acting beta agonists will not be excluded.
* 20. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure according to New York Heart Association Functional Classification ≥ 3, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring adverse events from TAB004, or compromise the ability of the subject to give written informed consent.
* 21. Untreated central nervous system and leptomeningeal metastases or requiring ongoing treatment for these metastases, including corticosteroids. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 28 days prior to study entry, have no evidence of new or enlarging metastases, and are off steroids.
* 22. Receipt of live attenuated vaccination within 28 days prior to study entry or within 30 days of receiving TAB004.
* 23. Any condition or treatment or diagnostic test that, in the opinion of the investigator or sponsor, would interfere with evaluation of TAB004 or interpretation of subject safety or study results.
* 24. Pregnancy or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by RECIST 1.1 | 2 years
  ORR
Duration of Response (DOR) by RECIST 1.1 | 2 years
  DOR
Disease Control Rate (DCR) by RECIST 1.1 | 2 years
  DCR
Time to response (TTR) by RECIST 1.1 | 2 years
  TTR
Progression-free survival (PFS) by RECIST 1.1 | 2 years
  PFS
Overall survival (OS) by RECIST 1.1 | 2 years
  OS
BTLA receptor occupancy (RO) of blood | 2 years
  RO
Maximum Plasma Concentration (Cmax) after single dose injection of TAB004 and for toripalimab | 2 years
  Cmax
Peak Time (Tmax) after single dose injection of TAB004 and for toripalimab | 2 years
  Tmax
Area Under the Curve (AUC) after single dose injection of TAB004 and for toripalimab | 2 years
  AUC
t1/2 after single dose injection of TAB004 and for toripalimab | 2 years
  t1/2 half life
Plasma clearance (CL) after single dose injection of TAB004 and for toripalimab | 2 years
  Plasma clearance (CL)
Apparent volume of distribution (V) after single dose injection of TAB004 and for toripalimab | 2 years
  volume of distribution (V)
Minimum Plasma Concentration (Cmin) of steady state after multiple dose injection of TAB004 and for toripalimab | 2 years
  Cmin
Apparent volume of distribution of steady state (Vss) after multiple dose injection of TAB004 and for toripalimab | 2 years
  volume of distribution of steady state (Vss)
The presence of anti-drug antibody (ADA) after multiple dose injection of TAB004 and for toripalimab | 2 years
  ADA
Accumulation after multiple dose in injection of TAB004 and for toripalimab | 2 years
  Accumulation

OTHER OUTCOMES:
Correlation analysis of HVEM expression of tumor and ORR | 3 years
  BTLA ligand expression with ORR, PD-L1 expression with ORR
Correlation analysis of HVEM expression of tumor and DCR | 3 years
  BTLA ligand expression with DCR,PD-L1 expression with DCR
Correlation analysis of HVEM expression of tumor and PFS | 3 years
  BTLA ligand expression with PFS, PD-L1 expression with PFS
Correlation analysis of HVEM expression of tumor and OS | 3 years
  BTLA ligand expression with OS, PD-L1 expression with OS

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yao, PhD, Study Director — TopAlliance Biosciences, Inc.
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona College of Medicine-Tucson, Tucson, Arizona
  - UCLA Health Westwood Cancer Care, Los Angeles, California
  - University of California Irvine (UCI) Medical Center, Orange, California
  - University of California San Francisco (UCSF) Medical Center-Mission Bay, San Francisco, California
  - University of California at San Francisio, San Francisco, California
  - Boca Raton Clinical Research (BRCR), Boca Raton, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - University of Iowa Hospitals, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Northwell Health, New Hyde Park, New York
  - New York Presbyterian / Weill Cornell Medical Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - UC Health - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin